CLINICAL TRIAL: NCT04729946
Title: Clinical and Urgent Colonoscopy Outcomes Using the Pure-Vu® Cleansing System in Hospitalized Patients With Lower Gastrointestinal Bleeding: A Single-Center Prospective Pilot Study
Brief Title: Clinical and Urgent Colonoscopy Outcomes Using the Pure-Vu® Cleansing System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: The Cleveland Clinic (Other)
Collaborators: Motus GI Medical Technologies Ltd (Industry)
Responsible Party: Principal Investigator, Brian Baggott, Vice Chair, Operations, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20-884
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Lower Gastrointestinal Bleeding; Hemostatic Disorder
Keywords: Colonoscopy; Bowel Preparation
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Single-Center Pilot Study
Masking Description: No Masking is planned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pure-Vu Treatment (Experimental): Participants in this arm will undergo colonoscopy using the Pure-Vu cleansing device.
  Interventions: Device: Pure-Vu Cleansing Device

INTERVENTIONS:
Device: Pure-Vu Cleansing Device — The Pure-Vu device attaches to the colonoscope and provides colonic cleansing during urgent colonoscopy without the need for a bowel preparation

SUMMARY:
The Pure-Vu® System can be effectively used as a cleansing device in patients admitted with acute LGIB to the intensive care unit and the regular nurse floor (RNF) bypassing the need to administer an oral bowel preparation for adequate visualization and hence decreasing time to colonoscopy and improving diagnostic and therapeutic yield.

DETAILED DESCRIPTION:
Acute lower gastrointestinal bleeding (LGIB), while generally defined as gastrointestinal bleeding distal to the ligament of Treitz, can be categorized into small bowel and colorectal bleeding, two sites with distinct presentations as well as diagnostic and management options (1). Acute LGIB secondary to a colorectal source usually presents with sudden onset hematochezia with or without acute blood loss anemia and hemodynamic instability, and usually leads to multiple invasive procedures and hospitalizations. It accounts for up to one-third of all hospitalizations related to GIB (2). The current guidelines recommend urgent colonoscopy to be performed within 8 to 24 hours of presentation and after adequate colon preparation to improve visualization and diagnostic/therapeutic yield (1). While studies looking at optimal timing of colonoscopy are limited for patients with acute LGIB, a study comparing 48 patients with diverticular bleeding who underwent colonoscopy after rapid polyethylene glycol (PEG) preparation and within 12 hours of presentation with endoscopic hemostasis compared to 73 controls without endoscopic hemostasis, found a significant improvement in outcomes in the group that underwent hemostasis, including bleeding (0% vs. 53%) and hospital length (median of 2 days vs. 5 days) (3). In another RCT of 100 patients presenting with LGIB, colonoscopy within 8 hours of presentation after rapid preparation lead to a more definite diagnosis compared to patients who underwent elective colonoscopy within 96 hours of presentation (4). Urgent colonoscopy however requires the rapid administration of a large volume bowel preparation over 3-4 hours until the rectal effluent is clear (1). Purge preparation can be challenging in critically ill patients and frequently requires the placement of a nasogastric tube for administration of the preparation which could place the patient at risk of aspiration, poor tolerance, and rarely, electrolyte imbalances (1). Moreover, bleeding can subside while awaiting resuscitation and bowel preparation prior to endoscopic intervention, which could lead to a decreased diagnostic and therapeutic yield. The guidelines recommend against unprepped colonoscopy due to poor visualization and increased perforation risk (1). A pilot study looked at the effect of "hydroflush colonoscopy" in acute LGIB with minimally prepped colons (tap water enema without oral preparation). "Hydroflush colonoscopy" was defined as colonoscopy using a combination of a water jet pump irrigation and a mechanical endoscope suction device (BioVac direct suction device). Out of the 12 patients included, the cecum was reached 69% of the time and endoscopic visualization was found to be adequate to find the source of bleeding in all procedures (5). The Pure-Vu® System (MotusGI Ltd.), a novel Food and Drug Administration (FDA) 510k cleared intra-procedural cleansing device, has been recently introduced. The Pure-Vu® System integrates with the colonoscope and generates a pulsed vortex mixture of water and air in order to remove debris and is active at the time of cleansing to evacuate colonic contents simultaneously (6). Its effectiveness has been studied in colonoscopies requiring minimal preparation regimens with excellent and safe results (7,8). A multicenter European feasibility study looked at 47 patients referred for colonoscopy who received a limited bowel preparation and found significant improvement in the proportion of patients with adequate preparation, with a median Boston bowel preparation score (BBPS) increased from 3[0-5] to 9 [8-9] (8). The REDUCE trial (9), another multicenter, single-arm study, was the first trial to study Pure-Vu® in the inpatient setting, which enrolled 95 hospitalized subjects. Adequate bowel preparation improved from 38% (95% CI 28,49) to 96% (CI 90-99) in the evaluated segments. The mean BBPS improved from 1.74 in the left colon, 1.74 in the transverse colon, 1.5 in the right colon to 2.89, 2.91 and 2.86 respectively (p<0.001) (9).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients in the ICU or the RNF with acute LGIB (defined as maroon-colored stool or bright red blood per rectum with suspicion of acute blood loss anemia, and hemodynamically stable and/or stabilized at the time of procedure . Hospitalized patients include:

  * Patients who develop LGIB while admitted for different reasons
  * Patients transferred from an outside hospital for further management of acute LGIB
  * Patients admitted through the emergency room for management of acute LGIB
* At least 22 years old
* Undergoing urgent colonoscopy under monitored anesthesia care or conscious sedation

Exclusion Criteria:

* Suspicion for bowel obstruction/ stricture
* Toxic megacolon or severe colitis (determined by degree of colitis on imaging and clinical condition including pain, fevers, abdominal exam, elevated inflammatory markers)
* Active Diverticulitis

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Adequate Bowel Preparation | During the colonoscopy procedure, typically less than 1 hour
  The proportion of participants who achieve an adequate bowel preparation to identify bleeding lesions

SECONDARY OUTCOMES:
Diagnostic yield | During the colonoscopy procedure, typically less than 1 hour
  The frequency with which investigators are able to successfully identify the source of bleeding.
Therapeutic Yield | During the colonoscopy procedure, typically less than 1 hour
  The frequency with which investigators are able to successfully control bleeding through endoscopic intervention
Re-bleeding rate | 48 hours post-colonoscopy
  The proportion of participants who experience recurrence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Brian Baggott, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04729946/Prot_000.pdf
  • Informed Consent Form (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT04729946/ICF_001.pdf